CLINICAL TRIAL: NCT02675283
Title: Case Finding for Coeliac Disease Using a Point of Care Test in a Pharmacy Setting: A Feasibility Study
Brief Title: Case Finding for Coeliac Disease Using a Point of Care Test in a Pharmacy Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH19172
Record Dates: First submitted 2016-01-25; First posted 2016-02-05 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Coeliac Disease
Keywords: Point of care test; Diagnosis; Case finding
MeSH Terms: conditions — Celiac Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- coeliac disease point of care test (Other): Patients will be consented for a finger prick point of care test, Simtomax, at the pharmacy.
  Interventions: Device: Simtomax

INTERVENTIONS:
Device: Simtomax — Patients will undertake a finger prick point of care test, Simtomax, at the pharmacy. A sample of 25 μl of capillary venous blood is required which can be obtained through a simple finger prick technique. The sample is then applied to the test device, followed by the application of 5 drops of the provided buffer solution. The result can be read after 10 minutes. Positive results are indicated by the presence of a solid red line, with a single line for a combined IgA and IgG DGP positivity, and a single line for the presence of total IgA. An in-built control line ensures a correctly functioning test.
  Other Names: Point of care test

SUMMARY:
This study aims to assess whether it is feasible to use a point of care test to increase the detection of coeliac disease in a pharmacy setting.

DETAILED DESCRIPTION:
Coeliac disease (CD) is an autoimmune condition characterised by mucosal damage of the small intestine by dietary gluten. CD affects 1 in 100 people. However, patients do not always have symptoms, resulting in 5 undiagnosed patients to every known case of CD. Undiagnosed CD can lead to complications such as vitamin and mineral deficiencies, osteoporosis and small bowel lymphoma, as well as impairing quality of life.

Currently, patients are diagnosed with a conventional blood test for coeliac antibodies (anti-TTG) as a first line test. Simtomax®, a new coeliac point of care test (POCT), has become available. It is a finger prick test that provides results of a coeliac antibody, deaminated gliadin peptide, within 10 minutes. Studies showed that Simtomax is as accurate as anti-TTG, with a 92.7% chance of detecting CD and 98.7% chance of ruling out CD.

This study aims to assess whether the POCT can increase the detection of adult coeliac disease when used in a pharmacy setting. A feasibility study using a case-finding approach will be conducted at 5 pharmacies in Sheffield over 20 months. It will be funded by Professor Sanders' research funds.

Customers who enter the pharmacies will be approached by the principal investigator (PI). Eligible participants (those with symptoms suggestive of or risk factors for CD) will be consented for the POCT by the PI. The POCT will be carried out at the pharmacies. Any participant with a positive test will be advised to see his GP to be referred for a gastroscopy at the Royal Hallamshire Hospital to confirm the diagnosis. Once diagnosed, the participant will follow the standard management pathway for any patients with CD.

Results of the study will be compared to the established prevalence of CD of 1%, to assess whether using POCT in a pharmacy setting can increase the detection of adult CD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over, and
2. Purchasing gastrointestinal medications, including:

   * Over the counter medications (i.e. medicines purchasable without a prescription or supervision of a pharmacist)
   * Pharmacy medications (i.e. medicines purchasable from a pharmacy without a prescription but provided under the supervision of a pharmacist. These medicines are kept 'behind the counter' and are not available on the pharmacy shelves.)
   * Prescription only medications (i.e. medicines only available with a prescription that is issued by a GP or another suitably qualified healthcare professional), and/ or
3. Suffering from any of the following:

   * Persistent unexplained abdominal or gastrointestinal symptoms
   * Prolonged fatigue
   * Unexpected weight loss
   * Severe or persistent mouth ulcers
   * Unexplained iron, vitamin B12 or folate deficiency
   * Type 1 diabetes
   * Autoimmune thyroid disease
   * Irritable bowel syndrome
   * Metabolic bone disorder (reduced bone mineral density or osteomalacia)
   * Unexplained neurological symptoms (particularly peripheral neuropathy or ataxia)
   * Unexplained subfertility or recurrent miscarriage
   * Persistently raised liver enzymes
   * Dental enamel defects, and/ or 4 Have first degree relatives with coeliac disease

Exclusion Criteria:

* previous diagnosis of coeliac disease, or
* previous or current investigation for coeliac disease.
* age under 18.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The prevalence of CD in this study cohort as a result of a case finding approach using a POCT in a pharmacy setting. | Baseline - 20 months
  This feasibility study will describe the prevalence of CD in this study cohort. This will be compared to the established prevalence of CD of 1% in the general population.

SECONDARY OUTCOMES:
The proportion of individuals agreeing to fill in the eligibility questionnaire. | Baseline - 20 months
The proportion of individuals undertaking the POCT. | Baseline - 20 months
The proportion of individuals undergoing a gastroscopy with duodenal biopsies. | Baseline - 20 months

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No